CLINICAL TRIAL: NCT06665087
Title: Comprehensive Geriatric Assessment (CGA) Guided Ultrafractionated Radiotherapy and First-line Systemic Treatment in Elderly or Frail Patients with Metastatic Colorectal Cancer
Brief Title: CGA Guided Ultrafractionated RT and First-line Systemic Treatment in Elderly or Frail Patients with MCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-157-3710
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — spartalizumab; Drug Therapy; Fluorouracil; raltitrexed; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGA cohort (Experimental): all patients will receive Ultrafractionated Radiotherapy (RT) and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment. All patients will receive Ultrafractionated RT and PD-1 antibody. Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed, with/without targeted therapy, and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, with/without targeted therapy, and BSC.
  Interventions: Drug: Ultrafractionated RT and CGA Guided systemic treatment.; Radiation: Ultrafractionated Radiotherapy; Drug: PD-1 antibody; Drug: Chemotherapy (Fluorouracil); Drug: Chemotherapy (Raltitrexed); Drug: Chemotherapy (Oxaliplatin); Drug: Chemotherapy (CPT-11); Drug: Targeted Therapy (anti-VEGF); Drug: Targeted Therapy (anti-EGFR)
- external control cohort (Other): external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.
  Interventions: Drug: Chemotherapy (Fluorouracil); Drug: Chemotherapy (Raltitrexed); Drug: Chemotherapy (Oxaliplatin); Drug: Chemotherapy (CPT-11); Drug: Targeted Therapy (anti-VEGF); Drug: Targeted Therapy (anti-EGFR)

INTERVENTIONS:
Drug: Ultrafractionated RT and CGA Guided systemic treatment. — in cohort 1, all patients will receive Ultrafractionated RT (1Fx every 3 or 4weeks) and Sintilimab (q3w). Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed, with/without targeted therapy, and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, with/without targeted therapy, and BSC.
  Arms: CGA cohort
Radiation: Ultrafractionated Radiotherapy — 1Fx every 3 or 4weeks
  Arms: CGA cohort
Drug: PD-1 antibody — Sintilimab
  Arms: CGA cohort
Drug: Chemotherapy (Fluorouracil) — 5-Fluorouracil or capecitabine
Drug: Chemotherapy (Raltitrexed) — Raltitrexed
Drug: Chemotherapy (Oxaliplatin) — Oxaliplatin
Drug: Chemotherapy (CPT-11) — Irinotecan
Drug: Targeted Therapy (anti-VEGF) — anti-VEGF antibody
Drug: Targeted Therapy (anti-EGFR) — anti-EGFR antibody

SUMMARY:
This is a prospective, multicentre, cohort study. For cohort 1(CGA cohort), experimental cohort, older or Frail patients with metastatic colorectal cancer will receive Ultrafractionated Radiotherapy (RT) and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment. All patients will receive Ultrafractionated RT and PD-1 antibody. Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive single agent chemotherapy, with/without targeted therapy, and BSC; Fit patients will receive doublet chemotherapy, with/without targeted therapy, and BSC.

For cohort 2 (external control cohort), external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.

The primary endpoint is Progression Free Survival (PFS). The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, quality of life (QoL), the Overall Response Rate (ORR), 1-year Disease-specific survival (DSS) rate, 1-year overall survival (OS) rate etc.

DETAILED DESCRIPTION:
This is a prospective, multicentre, cohort study. For cohort 1(CGA cohort), experimental cohort, older or Frail patients with metastatic colorectal cancer will receive Ultrafractionated Radiotherapy (RT) and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment. All patients will receive Ultrafractionated RT and PD-1 antibody. Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed, with/without targeted therapy, and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, with/without targeted therapy, and BSC.

For cohort 2 (external control cohort), external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.

The primary endpoint is Progression Free Survival (PFS). The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, quality of life (QoL), the Overall Response Rate (ORR), 1-year Disease-specific survival (DSS) rate, 1-year overall survival (OS) rate etc.

ELIGIBILITY:
Inclusion Criteria:

1. ≥70y, or, ≥60 and <70y but ECOG≥2;
2. male or female;
3. metastatic colorectal cancer;
4. at least one measurable leasion;
5. the primary lesion could be 1)previously resected, or 2) not resected or recurred, and not been previously irradiated;
6. no more than 10 lesions, and all the lesions could be safely irradiated.
7. life expectancy is more than 3 months;
8. no previous standard first-line anti-cancer treatment(including 5-FU/ Capecitabine/Raltitrexed, oxaliplatin, or irinotecan), or more than 6 months after perioperative chemotherapy;
9. No immunotherapy prior to enrollment;
10. With good compliance during the study;
11. Signed written informed consent.

Exclusion Criteria:

1. Known history of other malignancies within 3 years，except cured skin cancer, cervical cancer in situ, thyroid carcinoma, or clinical controlled prostate cancer;
2. Individuals with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorders that, in the judgment of the investigator, are of such clinical severity that they may prevent the signing of an informed consent form or affect the patient's adherence to oral medications;
3. Individuals with clinically serious (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmia requiring pharmacologic intervention, or history of myocardial infarction within the last 12 months;
4. Individuals with a history of organ transplantation requiring immunosuppressive therapy and long-term hormone therapy;
5. Individuals with autoimmune diseases;
6. Individuals with severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
7. Baseline hematology and biochemistry did not meet the following criteria: Hb≥80g/L; NEU ≥1.5×109/L; PLT ≥100×109/L（PLT ≥80×109/L if there were liver metastasis）; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; TB <1.5 times the upper limit of normal; Cr <1 time the upper limit of normal; Alb ≥30g/L;
8. Individuals allergic to any drug component of the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From the start of treatment until 3 months after the completion of therapy.
  Rate of chemotherapy, radiotherapy, targeted therapy, and immunotherapy related adverse events.
the Overall Response Rate (ORR) | up to 1 year since the start of treatment.
  the percentage of patients with a best overall response of complete response or partial response.
health-related quality of life (HRQOL) | baseline, and at 3, 6 and 12 months.
  EORTC QLQ C30 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core with 30 items] will be filled by all patients. Scores at different time points after treatment will be compared to baseline scores.
health-related quality of life (HRQOL) | baseline, and at 3, 6 and 12 months.
  EORTC QLQ CR29 [The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items] will be filled out by all patients. Scores at different time points after treatment will be compared to baseline scores.
1-year Disease-specific survival (DSS) rate | From the start of treatment until the date of death from the specific disease, assessed up to 12 months.
  rate of 1 year Disease-specific survival
1-year overall survival (OS) rate | From the start of treatment until the date of death from any cause, assessed up to 12 months.
  rate of 1 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhen ZHANG Principal Investigator, Principal Investigator — Fudan University